CLINICAL TRIAL: NCT00446069
Title: A Double-blind, Randomized, 2-way Cross-over, Phase II, Efficacy Trial in Cancer Patients to Assess the Overall Efficacy, Patient Preference, Morphine Related Side Effect Profile and Safety of the Egalet® Controlled Release Morphine Formulation 30-240 mg Once Daily Compared to MST Continus® 15-120 mg Twice Daily After 2 Weeks of Treatment
Brief Title: A Efficacy and Safety Trial of Controlled Release (CR) Morphine in Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Egalet Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MP-EG-002; EudraCT number: 2006-006579-19
Record Dates: First submitted 2007-03-09; First posted 2007-03-12 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Pain; Cancer
MeSH Terms: conditions — Pain; Neoplasms | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Egalet® morphine (Experimental)
  Interventions: Drug: Morphine Sulphate
- MST Continus® (Active Comparator)
  Interventions: Drug: Morphine Sulphate

INTERVENTIONS:
Drug: Morphine Sulphate — Egalet® morphine, Controlled Release 30 mg Oral tablet once daily for 2 weeks and MST Continus® 15 mg twice daily for 2 weeks

SUMMARY:
The purpose of the study is to determine the effect of Egalet® Morphine once daily compared to MST Continus twice daily on pain intensity and use of rescue medication for break through pain after 2 weeks of treatment in patients with pain due to cancer.

ELIGIBILITY:
Inclusion Criteria:

* The patient has stable strong opioid use equipotent to 30-240 mg oral morphine sulphate daily for a minimum of 2 weeks prior to entering the run-in phase.
* The patient has opioid-sensitive pain caused by active cancer.
* The patient is aged minimum 18 years.

Exclusion Criteria:

* The patient has a life expectancy less than 2 months.
* The patient has received chemotherapy or radiation therapy less than 4 weeks prior to entering run-in phase
* Patients with medical conditions contraindicating morphine treatment
* The patient has hepatic disease or impaired kidney function
* The patient is taking monoamine oxidase inhibitors (MAOIs) or has taken a MAOI within two weeks prior to entering baseline.
* The patient is taking other opioid agonists or antagonists, zidovudine or cimetidine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-08; Primary Completion 2008-06 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Use of rescue medication | 2 weeks treatment

SECONDARY OUTCOMES:
Pain intensity | 2 weeks treatment

CONTACTS AND LOCATIONS:
Overall Officials: Christine Andersen, MSc Pharm, Study Director — Egalet A/S
Locations (8):
- Lithuania (2):
  - Site 51, Kaunas
  - Site 50, Vilnius
- Poland (6):
  - Site 63, Bielsko-Biaia
  - Site 60, Bydgoszcz
  - Site 62, Poznan
  - Site 61, Warsaw
  - Site 64, Wroclaw
  - Site 65, Włocławek